CLINICAL TRIAL: NCT07172893
Title: A Non-Randomized Open Label Clinical Trial Evaluating the Efficacy, Safety, and Tolerability of DermaBind TL, a Placental Membrane Allograft Intended for Use in the Management of Non-Healing Ulcers
Brief Title: A Non-Randomized Open Label Clinical Trial Evaluating DermaBind TL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: HealthTech Wound Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTWCDBTL0001
Record Dates: First submitted 2025-07-18; First posted 2025-09-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcer (VLU)
Keywords: Placental allograft; Diabetic Foot Ulcer; Venous Leg Ulcer; DermaBind TL
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efficacy, Safety, and Tolerability of DermaBind TL (Experimental): The SOC therapy in this study is offloading of the DFU or VLU (Foot Defender® CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM Boot), appropriate sharp or surgical debridement, infection management and wound care covering with dehydrated Placental membrane tissue allograft (DERMABIND TL™), and a non-adherent dressing, followed by a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).
  Interventions: Biological: DermaBind TL

INTERVENTIONS:
Biological: DermaBind TL — Full-Thickness Dehydrated Placental Allograft

SUMMARY:
The purpose of this clinical evaluation is to collect patient outcome data and evaluate the efficacy, safety and tolerability of HealthTech DermaBind TL™ in patients with chronic non-healing wounds in patients with chronic non-healing ulcers.

DETAILED DESCRIPTION:
This clinical trial will assess the effectiveness of HealthTech Wound Care's medical intervention with the use of DermaBind TL™. HealthTech Wound Care will analyze data related to specific endpoints, such as, wound area preservation over time, rate of wound infection over time, rate of wound reoccurrence post-treatment through EOS, the average number of grafts used per subject and incidence of treatment-emergent adverse events. The goal is to determine whether the intervention produces the desired effects. HealthTech Wound Care will use each study subject's historical data in relation to existing treatments when summarizing data.

This study is a prospective, multi-center, open-label, single arm clinical trial designed to collect patient outcome data on commercially available dressing/covering for the protection of DFUs or VLUs over a 12-week treatment period. Wound assessment will be conducted by a clinician, Principal Investigator/Sub-Investigator at each site.

The study will include adult patients with chronic non-healing wounds that have failed to respond to standard or conservative treatments. These wounds may include diabetic foot ulcers and venous leg ulcers.

The treatment period will be 12 weeks, during which DermaBind TL™ will be applied to the affected wound. The study will monitor outcomes related to , wound area protection, infection rates, through EOS, and adverse events.

The study involves two phases: Screening and Treatment

ELIGIBILITY:
Inclusion Criteria:

* 1. Be an adult between 18 and 80 years of age at the time of consent 2. Presence of a DFU, Wagner Grade 1 or 2 (see Appendix A for definitions) on the plantar, lateral or dorsal aspect of the foot, extending through the dermis provided it is below the medial aspect of the malleolus.

  3. Subjects must have a diagnosis of Type I or Type II diabetes mellitus (DM) as defined by the American Diabetes Association
  1. for Type I DM, have been on a stable anti-diabetic treatment for at least 30 days before the baseline visit, or
  2. for Type II DM, must have been on a stable anti-diabetic medication for at least 30 days, or if diet-controlled only, must have been on stable diet-control for at least 6 months.

     4. For Type I and Type II DM, A1C must be equal or <10% in the last 30 days, or confirmed during the screening period (SV1 up to TV1) 5. Have a single target ulcer 6. If other DFU wounds are present on the same foot, they must be more than 2 cm distant from the index ulcer. [NOTE: If two or more DFUs are present with the same grade on the same foot, the index ulcer is the largest ulcer and the only one evaluated in the study.] 7. Have a wound with an area greater than 1cm2 and less than 25 cm2 and does not probe to bone 8. Index ulcer has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.

     9. Index ulcer must be a DFU with a Wagner Grade of 1 or 2. 10. Have an absence of infection based on the Infectious Disease Society of America criteria and as evidenced by radiographic evidence (X-ray, CT or MRI scan) performed during the 14 Screening Period (SV1-TV1). Radiological evidence must be completed, resulted and confirmed by the treating study physician prior to application of study graft to index ulcer.

     11. Have adequate circulation to the affected lower extremity confirmed during the screening period, defined as at least one of these criteria:

  <!-- -->

  1. TCOM ≥30 mmHg
  2. ABI between 0.7 and 1.3
  3. SPP >30 mmHg
  4. As an alternative, Arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle on the extremity the index ulcer is located.

     12. Have the ability to comply with protocol defined off-loading to the index ulcer and dressing change requirements 13. Patient is a non-tobacco user, including all forms of nicotine delivery (e.g., cigarettes, cigars, pipes, vaping devices, smokeless tobacco or nicotine patch) for a minimum of 4 weeks prior to the initial application of study graft. Verbal confirmation by subject is acceptable.

     14. Have the ability to understand the requirements of the study and to give informed consent 15. Have a life expectancy of greater than 6 months 16. Have failed conservative wound care treatment of the index ulcer for at least of 4 weeks 17. Patient will not require negative pressure therapy to the index ulcer, antimicrobial dressings, hyperbaric oxygen therapy to the index ulcer during the study period.

     18. Patient has not had radiation to the index ulcer site. 19. The index ulcer has a clean base, free of necrotic debris and infection at time of placement of treatment product.

     20. The index ulcer has been off-loaded, per protocol requirements, with a CAM boot (Foot Defender®) or TCC for a minimum of 14 days (+3 days) following SV1.

     21. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests at various timepoints during study participation.

     Exclusion Criteria:
* 1. Pregnant or lactating 2. Less than 18 years of age 3. Has continued tobacco use 4. Have a wound that decreased in size ≥30% between the Screening and Treatment Visits 5. Wound is showing signs of healing and that improvement is likely to continue without treatment (increased granulation, epithelization, decrease in size ≥ 30% reduction in wound surface area).

  6. Circulating hemoglobin A1c exceeding 10% within 30 days of the Screening Visit 7. Serum creatinine concentrations of 3.0 mg/dL or greater within 30 days prior to screening 8. The wound has been treated with biomedical or topical growth factors within the previous 30 days before the screening visit 9. Need for any additional concomitant dressing material other than the ones approved for this study 10. Osteomyelitis or bone infection of the affected foot as verified by x-ray or other radiographic modality within 30 days prior to the first screening visit. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).

  11. The inability to tolerate off-loading (a surgical shoe, removable cast walker or a total contact cast) 12. Have a known or suspected disease of the immune system 13. Have an active or untreated malignancy or active, uncontrolled connective tissue disease 14. Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.

  15. At the index ulcer site, presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement 16. Had undergone a revascularization procedure aimed at increasing blood flow in the treatment target limb less than 4 weeks before the baseline visit 17. Have serum aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels greater than three times the normal upper limit within 30 days prior to screening 18. Uncontrolled edema, lymphedema or venous HTN in the limb of the index ulcer 19. Undergone treatment to the index ulcer with a living skin equivalent within the last 4 weeks before screening 20. Undergone treatment to the index ulcer with a placental-derived allograft within the last 4 weeks before screening 21. Has the presence of any condition that in the opinion of the investigator places the subject at undue risk or potentially jeopardizes the quality of the data to be generated 22. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.

  23. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.

  24. Subjects with a previous diagnosis of HIV or Hepatitis C, regardless of current status .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-02-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Measure the protective effect of the wound covering on the wound over the 13-week treatment period | 13 weeks
  Size of wound will be measured using Clock method
  * 12 o'clock to 6 o'clock: Measure the length of the wound from the top (12 o'clock) to the bottom (6 o'clock).
  * 9 o'clock to 3 o'clock. Measure the width of the wound from the left (9 o'clock) to the right (3 o'clock).
  * Depth Measurement: Use a cotton tip applicator to measure the depth. Insert the applicator gently into the deepest part of the wound, mark the point where it meets the wound edge, and measure the length from the tip to the mark.
  * The area is then calculated as: Area (cm2) = Length (cm) × Width (cm), where length is the longest axis of the index ulcer and width is the longest orthogonal at an axis 90 degrees relative to the length.

SECONDARY OUTCOMES:
Preservation of the wound area over the study period | 13 Weeks
  Determination that the wound area does not increase through the 13 week study. This will be determined by the study physician and verified by an independent third party.
Monitor the rate of wound infection over the 13 week study | 13 Weeks
  Number of wound infections observed during 13 week study on the study wound. This will be determined by the study physician and verified by an independent third party.
Average number of DermaBind TL™ grafts used per subject | 13 Weeks
  Count the number of DermaBind TL grafts used per study subject to determine efficiency of use.
Incidence of treatment-emergent adverse events (TEAEs), including any clinically significant changes in vital signs, ankle-brachial index (ABI), and findings from physical exams, throughout the study period | 13 Weeks

OTHER OUTCOMES:
Product Wastage | 13 Weeks
  Total surface area of grafts used minus calculated surface area of index ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Stan Andrews, MS, Study Director — Professional Education and Research Institute
Locations (10):
- United States (10):
  - Midland Florida Clinical Research Center, DeLand, Florida
  - Pharmakon Medical Research, Palm Beach Gardens, Florida
  - Vital Medical Research, Sweetwater, Florida
  - EMbassy Research Network, Bloomfield Township, Michigan
  - US Foot and Ankle Specialists-Cary Satellite Site, Cary, North Carolina
  - US Foot and Ankle Specialists, Raleigh, North Carolina
  - US Foot and Ankle Specialists, Blue Ash, Ohio
  - Lower Extremity Institute for Research and Therapy, Boardman, Ohio
  - Perfizien Clinical Research, LLC., Houston, Texas
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: July 2026